CLINICAL TRIAL: NCT02824900
Title: Vibration Stimuli in Stroke Patients With Contraversive Pusher Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Nachum Soroker, MD (Other)
Collaborators: Tel Aviv University (Other)
Responsible Party: Sponsor-Investigator, Nachum Soroker, MD, head, Department of neurologic rehabilitation, Loewenstein rehabilitation hospital, Raanana,Israel, Loewenstein Hospital
Organization: Loewenstein Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: loe162315CTIL
Record Dates: First submitted 2016-06-29; First posted 2016-07-07 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-10

CONDITIONS: Stroke
Keywords: Vibration Stimuli; Contraversive Pusher Syndrome
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Vibration stimuli to neck (Experimental): Vibration stimuli to contralesional neck muscles, 5 days per week, for 2 weeks, 20 minutes per day + structured (conventional exercises) daily physiotherapy ~ 45 minutes.
  Interventions: Device: Vibration stimuli to neck muscles; Behavioral: conventional physiotherapy
- Vibration stimuli to hand (Active Comparator): Vibration stimuli to contralesional hand, 5 days per week, for 2 weeks, 20 minutes per day + structured (conventional exercises) daily physiotherapy ~ 45 minutes.
  Interventions: Device: Vibration stimuli to hand; Behavioral: conventional physiotherapy

INTERVENTIONS:
Device: Vibration stimuli to neck muscles
  Arms: Vibration stimuli to neck
Device: Vibration stimuli to hand
  Arms: Vibration stimuli to hand
Behavioral: conventional physiotherapy

SUMMARY:
The purpose of this study is to investigate the effects of vibration stimuli to contra lateral neck muscles on Contraversive Pusher Syndrome, function and neglect in stroke patients.

DETAILED DESCRIPTION:
12 post-stroke subjects will be recruited from neurological rehabilitation department at Loewenstein rehabilitation hospital, Raanana, Israel. The patients will be randomly assigned to one of two groups: 1) Experimental group. 2) Control group. The 2 weeks intervention (10 sessions) in each group will include vibration stimuli (frequency of 1 Hz and amplitude of 20 mm) for 20 minutes and structured standard physiotherapy for 45 minutes. The vibration stimuli in the experimental group will be done to the contralesional neck muscles, whereas the vibration stimuli in the control group will be done in the contralesional hand. Different assessments will be done before the intervention, after the first day of intervention, after two weeks of intervention and one months post-intervention. The tests will include: Clinical Scale for Contraversive Pushing, Lateropulsion Scale, Subjective Straight Ahead, Postural Assesment Scale for Stroke Patients, Anterior and Lateral Functional Reach Test, Posturography, Behavioral Inattention Test, Mesulam Cancellation Test, Line Bisection Test, Dynamic Starry Night and sensation.

Differences between groups will be calculated using t-tests or Mann-Whitney, depending on distribution of normality with corrections for multiple comparisons. Smallest Real Difference (SRD) will be calculated for detecting the minimal detectable change.

ELIGIBILITY:
Inclusion Criteria:

* First stroke
* Age 25-75 years
* Able to understand research instructions
* Stable clinical/metabolic state.
* Having Contraversive Pushing Syndrome, based on Clinical Scale for Contraversive Pushing.

Exclusion Criteria:

* Having previous neurological and orthopedic disability.
* Having pacemakers.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical Scale for Contraversive Pushing | Before the intervention, after the first day of intervention, after 2 weeks (end of intervention), and one month after the end of the intervention (follow up)
  Score range: 0-6. Score of zero indicates no pushing. Assesses pushing during spontaneous body posture, abduction and extension of the nonparetic extremities and resistance to passive correction of tilted posture.

SECONDARY OUTCOMES:
Change in Lateropulsion Scale | Before the intervention, after the first day of intervention, after 2 weeks (end of intervention), and one month after the end of the intervention (follow up)
  Score range: 0-17. Score of zero indicated no pushing. Assesses pushing during supine, sitting, standing, transfers and walking.
Change in Postural Assessment Scale for Stroke Patients | Before the intervention, after the first day of intervention, after 2 weeks (end of intervention), and one month after the end of the intervention (follow up)
  Score range: 0-36. Score of 36 indicates performance without help. Assesses maintenance and change of posture.
Change in Anterior and lateral functional reach test | Before the intervention, after the first day of intervention, after 2 weeks (end of intervention), and one month after the end of the intervention (follow up)
  Assesses equilibrium during sitting by measuring the distance of the anterior and lateral reaching with the upper limb.
Change in Posturography | Before the intervention, after the first day of intervention, after 2 weeks (end of intervention), and one month after the end of the intervention (follow up)
  Force Platform that calculates the amount of weight bearing on right and left side during sitting.
Change in Neglect - Behavioral Inattention Test | Before the intervention, after the first day of intervention, after 2 weeks (end of intervention), and one month after the end of the intervention (follow up)
  Score range: 0-146. Cutoff score: 129. Assesses the amount of attention to the left side during different task (such as: star and lines cancellation).
Change in Neglect - Mesulam Cancellation Test | Before the intervention, after the first day of intervention, after 2 weeks (end of intervention), and one month after the end of the intervention (follow up)
  Cancellation of forms. Assesses the amount of attention to the left side.
Change in Neglect - Line Bisection | Before the intervention, after the first day of intervention, after 2 weeks (end of intervention), and one month after the end of the intervention (follow up)
  Assesses the amount of deviation from the center of different lines decided by the subject. Assesses the amount of attention to the left side.
Change in Neglect - Test Dynamic Starry Night | Before the intervention, after the first day of intervention, after 2 weeks (end of intervention), and one month after the end of the intervention (follow up)
  Computerized task. Measures the reaction time and the number of neglected goals.
Change in Subjective Straight Ahead | Before the intervention, after the first day of intervention, after 2 weeks (end of intervention), and one month after the end of the intervention (follow up)
  Assesses the subjective alignment of the body.
Change in Sensory evaluation | Before the intervention, after the first day of intervention, after 2 weeks (end of intervention), and one month after the end of the intervention (follow up)
  Assesses superficial sensation in foot and proprioception in toes.

CONTACTS AND LOCATIONS:
Overall Officials: Sivi Frenkel-Toledo, PhD, Study Director — Loewenstein Hospital